CLINICAL TRIAL: NCT03807531
Title: A Non-randomized Trial of the Temporary Spur Stent System for the Treatment of Lesions Located in the Infrapopliteal Arteries Outside of the United States
Brief Title: A Study of the Temporary Spur Stent for the Treatment of Narrowing and Blockages in the Arteries Below the Knee
Acronym: DEEPER OUS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ReFlow Medical, Inc. (Industry)
Collaborators: ClinLogix. LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-002
Record Dates: First submitted 2019-01-11; First posted 2019-01-17 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Intervention Model Description: Multicenter, non-randomized, single-arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with TSS (Other): This is a single-arm study. Participating subjects will be treated with the Temporary Spur Stent System (TSS)
  Interventions: Device: Temporary Spur Stent System

INTERVENTIONS:
Device: Temporary Spur Stent System — Participating subjects that meet inclusion and exclusion criteria will undergo treatment of infrapopliteal occlusions and stenoses with the Temporary Spur Stent System according to protocol guidelines
  Other Names: G2-SPUR04X60, G2-SPUR03X60, G2-SPUR02x60

SUMMARY:
The purpose of this study is to evaluate the performance and safety of the Temporary Spur Stent System (TSS). The TSS is intended for use in conjunction with a commercially available drug coated balloon in the infrapopliteal arteries for the treatment of de novo or restenotic lesions.

This study is a prospective, non-randomized, multicenter, single arm trial, with sites in New Zealand, Germany, and Switzerland.

At least two and no more than 10 sites are expected to participate, with 100 subjects enrolled (no more than 40 at a single site).

The study follow up will take place over a period of 365 days. A vessel recoil substudy will be included for a select group of subjects.

DETAILED DESCRIPTION:
The purpose of this clinical study is to evaluate the performance and safety of the Temporary Spur Stent System (TSS) for subjects with infrapopliteal arterial disease.

The Temporary Spur Stent System is intended for use in conjunction with a commercially available drug coated balloon in the infrapopliteal arteries for the treatment of de novo or restenotic lesions.

The TSS has been developed to provide another treatment option for patients with Peripheral Arterial Disease (PAD), and Critical Limb Ischemia (CLI).

Up to 100 subjects will be treated with the Temporary Spur Stent System in conjunction with an approved Drug Coated Balloon (DCB). No less than 1 subject and no more than 40 subjects will be enrolled at a single site.

A vessel recoil substudy is included in the trial. The purpose of this study is to evaluate vessel recoil in a select group of subjects (no more than 10 per site, up to 35 subjects in total). This will be conducted by obtaining measurements using Optical Coherence Tomography (OCT), Intravascular Ultrasound (IVUS), or Quantitative Vascular Analysis (QVA) of the target vessel during the index procedure.

The statistical analysis for this trial will use as a comparator a performance goal derived from a meta-analysis of infrapopliteal balloon angioplasty. Descriptive statistics may be used to describe other data points.

Subjects will be asked to participate in a baseline evaluation visit, the index procedure, a 30 day follow up visit, a 90 day follow up visit, a 180 day follow up visit, and a 365 day follow up visit. The baseline evaluation and index procedure visits may be combined. At each follow up visit, the subject will undergo a physical exam with wound evaluation (if applicable) including pictures, a medication history and compliance review, Ankle Brachial and Toe Brachial Indices (ABI and TBI), a duplex ultrasound of the treated limb, review of symptoms, and Adverse Events (AE) assessment. Subjects may choose to withdraw from the study at any time, for any reason. If subjects choose to withdraw, they will be asked to undergo an unscheduled study visit consisting of the aforementioned procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is willing and able to provide informed consent and able to comply with the study protocol.
2. Life expectancy >1 year in the investigator's opinion
3. Subject is > 18 years of age.
4. Subject is Rutherford class 3-5.
5. Stenotic, restenotic, or occlusive lesions located in the infrapopliteal vessels, with target lesion that can be successfully crossed with a guidewire.
6. Target lesion must meet lesion-specific criteria in pre-screening by angiography (pre-screening with CTA, MRA or selective angiography may be performed prior to the index procedure)
7. Target vessel(s) reconstitutes(s) at or above the medial malleolus, with the target treated segment extending no more than 10 mm beyond the medial malleolus.

   Note: If the anterior tibial or posterior tibial arteries are treated, there must be inline flow to the foot.

   If the peroneal artery is treated, there must be at least one collateral supplying the foot.
8. Target lesion must begin no higher than the tibioperoneal trifurcation (popliteal arteries excluded).
9. Target vessel reference diameter is measured to be between 2.0 mm to 4.5 mm in diameter, assessed by one of the following methods after successful completion of guidewire crossing of the lesion site:

   1. Intravascular Ultrasound (IVUS)
   2. Optical Coherence Tomography (OCT)
   3. Quantitative Vascular Angiography (QVA).
10. Lesion length must be > 30 mm and < 150 mm.
11. Only one limb may be enrolled per subject. Up to two vessels may be treated per subject; if required, a second modality may be used for treatment in the non-target infrapopliteal vessel. Any treatment of the non-index vessel must be performed prior to the use of the investigative device and only one artery may be treated with the investigative device
12. The total treated segment is defined as the total length of artery treated with the investigational device. Target treatment length is <240 mm with a maximum segment of 150 mm separated by 30 mm of healthy tissue between treated lesions.
13. Successful pre-dilatation of the target lesion as outlined in the procedure instructions, defined as resulting in stenosis <50%, without resulting flow limiting dissection (Type D or greater), thrombus, or aneurysm by angiography prior to the insertion of the investigative device.
14. Iliac, SFA and popliteal inflow lesions can be treated using standard angioplasty and/or an approved stent (no atherectomy) during the index procedure or >30 days prior. Inflow lesions treated intraprocedure must be treated first, prior to consideration of treatment of infrapopliteal lesions. If pre-screening with angiography, CTA, MRA, or ultrasound has been performed <365 days prior to the procedure, intra-procedure angiography of the aorto-iliac vasculature is not required, however, the infrainguinal inflow must still be imaged using angiography during the index procedure. Inflow lesions must have a healthy vessel segment of >30 mm between the study lesion and the treated segment, defined as less than 50% stenosis without aneurysmal segments.
15. Retrograde access (in the infrapopliteal arteries) is permitted for lesion crossing, however, the Temporary Spur Stent System must be deployed from antegrade access
16. For subjects with bilateral disease, planned treatment of the contralateral limb must either be performed >30 days prior to the index procedure or > 14 days following the index procedure.

Exclusion Criteria:

1. Subject unwilling or unlikely to comply with the appropriate follow up time for the duration of the study in the opinion of the investigator.
2. Subject is pregnant or planning to become pregnant during the course of the trial.
3. Subject has an active infection that is not controlled at the time of the procedure, including septicemia or bacteremia.
4. Subject has osteomyelitis or a heel wound.
5. Planned major (above the ankle) amputation of the target limb. A planned or previous minor (transmetatarsal or digit amputation) is permitted
6. Recent myocardial infarction or stroke < 90 days prior to the index procedure.
7. Heart failure with Ejection Fraction < 35%
8. Impaired renal function (eGFR <25 mL/min) within 30 days of procedure and subjects on dialysis
9. Subject with vasculitis, systemic Lupus Erythematosus or Polymyalgia Rheumatica.
10. Subject receiving chronic or intravenous corticosteroid therapy.
11. Inability to tolerate dual antiplatelet and oral anticoagulation therapy.
12. Known allergies or sensitivities to heparin, antiplatelet, or other anticoagulant therapies which could not be substituted, and/or paclitaxel or an allergy to contrast media that cannot be adequately pre-treated prior to the index procedure.
13. The subject is currently enrolled in another investigational device or drug trial that may interfere with the endpoints of this study.
14. Known allergy to nitinol or nickel.
15. Prior stent(s) within the target vessel, or bypass surgery of or within the target vessel(s)
16. Target lesion is located within an aneurysm or associated with an aneurysm in the vessel segment either proximal or distal to the target lesion. Inflow must also be free of aneurysmal segments.
17. Previous treatment failure of inflow arteries (Iliac, SFA and popliteal) which required a surgical procedure. Prior bypass above the level of the infrapopliteal arteries is permitted.
18. Previous treatment of inflow lesions, if not treated during the index procedure, must have been performed >30 days prior to the index procedure.
19. Previous treatment of the target vessel <30 days prior to index procedure
20. Angiographic evidence of thrombus within target limb.
21. Inability to obtain antegrade access in the limb from which the investigative device can be deployed.
22. Extremely severe calcification classified as grade 4 as measured by the Peripheral Academic Research Consortium (PARC) score or the Peripheral Arterial Calcium Scoring System (PACSS) that, in the investigator's opinion, would not be amenable to PTA.
23. Type D dissections or greater incurred during pre-dilation or CTO crossing.
24. Significant (>50%) stenosis of inflow arteries or unsuccessful treatment of inflow lesions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-07-11 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Primary patency of treated lesion sites by duplex ultrasound in subjects who are free from clinically driven TLR (target lesion revascularization) | 6 months
  The primary performance endpoint will be primary patency of treated lesion sites by duplex ultrasound in subjects who are free from clinically driven TLR (target lesion revascularization).
Freedom from device and procedure-related death through 30 days post-procedure | 30 days
  The primary safety endpoint is freedom from device and procedure-related death through 30 days post-procedure

SECONDARY OUTCOMES:
Freedom from clinically driven target lesion revascularization through 6 months post procedure. | 6 months
  The secondary efficacy endpoint is freedom from clinically driven target lesion revascularization through 6 months post procedure.
Decrease in Rutherford class score at 3, 6 and 12 months. | 3, 6, and 12 months
  The second secondary efficacy measurement is decrease in Rutherford class score at 3, 6 and 12 months. Rutherford score is a classification system for patients with peripheral vascular disease.
  Categories are numbered from 0 to 6, with 0 being asymptomatic, and 6 being major tissue loss, functional foot no longer salvageable. Higher values are therefore considered a worse outcome.
  Rutherford class zero: No symptoms; Rutherford class 1: Mild Claudication (minimal leg pain with ambulation) symptoms; Rutherford Class 2: Moderate Claudication (moderate leg pain with ambulation); Rutherford Class 3: Severe claudication (severe leg pain with ambulation); Rutherford Class 4: Ischemic Rest pain (leg pain at rest); Rutherford Class 5: Minor tissue loss (nonhealing ulcer, focal gangrene, diffuse pedal ischemia); Rutherford class 6: Major tissue loss (extending above the transmetatarsal TM level, functional foot no longer salvageable.
Wound healing for subjects with Rutherford class 5 at 6 and 12 months, as assessed by the investigator using WIfI score and descriptive characteristics, including change in wound size measured by any decrease in wound surface area. | 6 and 12 months
  The third secondary efficacy endpoint is wound healing for subjects with Rutherford class 5 at 6 and 12 months, as assessed by the investigator using WIfI score and descriptive characteristics, including change in wound size measured by any decrease in wound surface area.
  The WIfI classification scoring system is a grading system using a composite score of wound (W), ischemia (I), and foot infection (fi). These three different categories are graded from 0 to 3 with 0 being the best and 3 being the worst.
  The total score will be provided (clinical stage 1-5), which is used to estimate the risk for major amputation at one year. Patients with a score of 1 are considered low risk, and patients with a score of 5 are considered high risk (foot not salvageable). Therefore, higher values are considered a worse outcome.
  The composite score is calculated by adding up the score from each category.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Holden, MBChB, Principal Investigator — Auckland Hospital
Locations (6):
- Germany (4):
  - Klinikum Hochsauerland Klinik für Angiologie, Arnsberg
  - Universitats Herzzentrum Bad Krozingen, Bad Krozingen
  - Universitätsklinikum Leipzig, Leipzig
  - RoMed Klinikum Rosenheim, Rosenheim
- Auckland City Hospital, Auckland, New Zealand
- Ospedale di Lugano Civico, Lugano, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mills JL Sr, Conte MS, Armstrong DG, Pomposelli FB, Schanzer A, Sidawy AN, Andros G; Society for Vascular Surgery Lower Extremity Guidelines Committee. The Society for Vascular Surgery Lower Extremity Threatened Limb Classification System: risk stratification based on wound, ischemia, and foot infection (WIfI). J Vasc Surg. 2014 Jan;59(1):220-34.e1-2. doi: 10.1016/j.jvs.2013.08.003. Epub 2013 Oct 12. PMID 24126108